CLINICAL TRIAL: NCT06965075
Title: ObeSity and Jobs in SoCioeconomically Disadvantaged CommUnities --The SCULPT-Job Study
Brief Title: The SCULPT-Job Cohort Study
Acronym: SCULPT-Job
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-26093 B
Record Dates: First submitted 2025-05-01; First posted 2025-05-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Weight Maintenance; Weight Loss; Stress, Psychological; Job Stress; Diabetes Prevention; Obesity; Cardiovascular Risk Factor; Cardiovascular Diseases
MeSH Terms: conditions — Weight Loss; Stress, Psychological; Occupational Stress; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes Prevention Program (Experimental): The DPP is a behavioral obesity and diabetes prevention program run by the YMCA, over a 12-month period.
  Interventions: Behavioral: Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — Diabetes Prevention Program (DPP) is a one-year lifestyle modification program that helps adults at risk for developing type 2 diabetes gain tools for healthy living.
  Other Names: DPP

SUMMARY:
This is an research study about clinical, psychosocial, and behavioral factors that impact weight loss, weight maintenance, and cardiovascular disease in socially disadvantaged persons.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of the Diabetes Prevention Program (DPP) at 12 months among socioeconomically diverse participants by examining: changes in body mass index (BMI); improvements in ideal cardiovascular health scores (based on AHA 2020 goals and Life's Essential 8, where sleep data is available); and reductions in psychosocial stress.

ELIGIBILITY:
Inclusion Criteria:

•. Inlcudes participants from socioeconomically diverse backgrounds, age > 18 years old, and BMI > 25 kg/m2 (for Asian ethnicity BMI> 22 kg/m2).

Exclusion criteria will include pregnancy or post-partum state (< 12 months post-partum), history of diabetes (type 1 or 2), history of myocardial infarction, stroke or cardiac arrest in the prior 2 years, history of physician diagnosed cognitive, developmental or psychiatric conditions, recent orthopedic diagnosis or surgery (< 6 months) , inability to speak English, Spanish, or Chinese, persons facing housing eviction or undergoing an active housing leasing process (e.g getting their credit report in shape for a potential lease, in the process of getting a new housing lease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
BMI Change | Baseline and 12 month
  Weight will be measured using a calibrated digital scale to the nearest 0.1 kg. Height will be measured using a stadiometer. Waist and hip measurements will be performed using vinyl retractable tape to the nearest 0.1 cm at the smallest horizontal portion of the waist (highest horizontal point of the iliac crest with minimal respiration) and largest area of the hip.
BMI Maintenance | Baseline and 12 month
  The primary analysis of the maintenance phase will include 18-month outcomes, allowing 0-to-12 and 12-to-18 month linear changes by study arm. This model will estimate and compare mean (95% CI) 0-to-18 month changes by study arm: under the hypothesis that differential changes through month 12 will be maintained over the following 6 months, 12- and 18-month differences (95% CI) between arms will be similar (i.e., same sample size calculation). For descriptive purposes, we will compare the later slopes to quantify differential recidivism; within-arm 95% CIs that exclude positive values will demonstrate maintenance of intervention-period weight loss
Ideal Cardiovascular Health | Baseline and 12 month
  AHA 2020 ideal cardiovascular health score will be used as an index about cardiovascular health consisting of health behaviors and factors. Ideal cardiovascular health is defined as: BMI < 25 kg/m2, > 150 min/week of moderate physical activity, a healthy diet pattern including sufficient amounts of fruits and vegetables, optimal blood pressure (< 120/<80 mmHg), fasting glucose (< 100 mg/dL), total cholesterol < 200, and never smoking or quit smoking for more than 12 months
  For analysis, the investigators will score each item-level category as (0,0.5,1), respectively. This step expands the granularity of ICH Scores from 8 to 15 values, allowing finer measure of longitudinal change during the intervention and maintenance periods. For descriptive purposes,the investigators will compare the later slopes to quantify differential recidivism; within-arm 95% CIs that exclude positive values will demonstrate maintenance of intervention-period weight loss.

SECONDARY OUTCOMES:
Cumulative Stress | Baseline and 12 month
  The construct "cumulative psychological stress"(CPS), will be used to capture eight types of stress that commonly affect individuals over a life-course. The stressors include negative and traumatic life events, work-family stress, work, financial stress, intimate partner stress, neighborhood stress, and everyday discrimination. The questionnaire was constructed using a battery of scales approach that utilizes scales that have good psychometric properties that were assembled for the Chicago Community Health Aging (CCAHS), American Changing Lives, and Alameda County and Detroit Area Studies. Weights were assigned to each of the 8 domains comprising the cumulative stress score based on the reciprocal of the standard deviation of the scores for questions in each domain. The 8 domain-specific weighted scores were then added to create the cumulative stress score (CPS; range 16-385), with higher values representing higher stress.
Impulsivity | Baseline and 12 month
  The following indicators will be obtained: Self-reported indicators of trait impulsivity via the Barratt Impulsiveness Scale.
Cellular Aging Biomarkers | Baseline and 12 month
  To measure the change in telomeres, telomere length processing will be performed using finger-stick blood samples collected from participants at baseline and 12 months. Approximately 30 microliters of blood will be collected.
  Relative mean telomere length will be measured from DNA by a quantitative polymerase chain reaction (qPCR) assay as (T)/(S) ratio. The inter-assay coefficient of variability for telomere length measurement is 3.7%. The intra-assay coefficient of variability is 2.5% (equivalent to 0.13 kilobases/baseline mean)
Binge Eating | Baseline and 12 month
  BIS captures impulsive decision making, lack of planning, and impaired attention. We will assess binge eating by evaluating binge eating frequency using the methods from the Framingham Heart Study and severity from a 16 item binge eating scale, BES.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Albert, MD, Principal Investigator — University of California, SF
Locations (1):
- YMCA-Bayview, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baranowski T, Cullen KW, Nicklas T, Thompson D, Baranowski J. Are current health behavioral change models helpful in guiding prevention of weight gain efforts? Obes Res. 2003 Oct;11 Suppl:23S-43S. doi: 10.1038/oby.2003.222. PMID 14569036
- [Background] Baum A, Garofalo JP, Yali AM. Socioeconomic status and chronic stress. Does stress account for SES effects on health? Ann N Y Acad Sci. 1999;896:131-44. doi: 10.1111/j.1749-6632.1999.tb08111.x. PMID 10681894
- [Background] Kumanyika SK, Whitt-Glover MC, Gary TL, Prewitt TE, Odoms-Young AM, Banks-Wallace J, Beech BM, Halbert CH, Karanja N, Lancaster KJ, Samuel-Hodge CD. Expanding the obesity research paradigm to reach African American communities. Prev Chronic Dis. 2007 Oct;4(4):A112. Epub 2007 Sep 15. PMID 17875256
- [Background] Lantz PM, House JS, Mero RP, Williams DR. Stress, life events, and socioeconomic disparities in health: results from the Americans' Changing Lives Study. J Health Soc Behav. 2005 Sep;46(3):274-88. doi: 10.1177/002214650504600305. PMID 16259149
- [Background] Spinella M. Normative data and a short form of the Barratt Impulsiveness Scale. Int J Neurosci. 2007 Mar;117(3):359-68. doi: 10.1080/00207450600588881. PMID 17365120
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Albert MA, Durazo EM, Slopen N, Zaslavsky AM, Buring JE, Silva T, Chasman D, Williams DR. Cumulative psychological stress and cardiovascular disease risk in middle aged and older women: Rationale, design, and baseline characteristics. Am Heart J. 2017 Oct;192:1-12. doi: 10.1016/j.ahj.2017.06.012. Epub 2017 Jun 28. PMID 28938955